CLINICAL TRIAL: NCT01963390
Title: Testosterone Therapy and Its Effects on Metabolic Function
Brief Title: Metabolomics During Testosterone Therapy
Status: Completed | Type: Observational
Sponsor: Men's Health Boston (Other)
Responsible Party: Sponsor
Other Study IDs: 2012P000184
Record Dates: First submitted 2013-10-13; First posted 2013-10-16 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Testosterone Deficiency
Keywords: Hypogonadism; Testosterone Deficiency
MeSH Terms: conditions — Hypogonadism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples obtained for metabolomics
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Testosterone therapy: The study population is a cohort of testosterone deficient men who are planning on undergoing testosterone therapy at an outpatient men's health clinic.
  Interventions: Drug: Testosterone Therapy

INTERVENTIONS:
Drug: Testosterone Therapy — In this observational study we will be enrolling testosterone deficient men who intend to undergo testosterone therapy.

SUMMARY:
One promising but understudied area in the field of testosterone (T) therapy is its effect on metabolism and the development of type II diabetes. Metabolomics is a powerful research tool that can detect very early signs of metabolic derangement that may lead to metabolic disease. In this observational study, investigators aim to apply metabolomics in order to better understand how T therapy influences metabolism. In a clinical population of outpatient men with T deficiency investigators will perform comprehensive clinical evaluations and also obtain blood for metabolomics. This will be done once prior to T therapy and again after 4-6 months of T therapy. Investigators hypothesize that they can detect metabolic derangements in men with T deficiency and that these derangements will improve with T therapy.

DETAILED DESCRIPTION:
One promising but understudied area in the field of T therapy is its effect on insulin resistance (IR) and the development of type II diabetes and cardiometabolic disease. Although several clinical studies suggest T therapy improves metabolic parameters and may prevent disease progression, a mechanism for understanding this process is lacking. Investigators propose to use metabolomics to shed light on how metabolic function changes with T therapy.

Metabolomics is an established investigative tool that measures hundreds of unique chemical markers (metabolites) involved in normal and diseased cellular processes from a blood sample. Previous studies using the Metabolite Profiling Platform at the Broad Institute of Harvard/Massachusetts Institute of Technology applied tandem liquid chromatography-mass spectrometry (LC-MS)-based metabolomics to large, population-based cohorts. These studies identified and validated highly sensitive signatures of IR that successfully predicted occult risk for type II diabetes in clinically normal men. Investigators now plan to apply metabolomics to a clinical population in order to obtain a new perspective on the biochemical metabolic changes that occur based on a man's testosterone status. Investigators plan to study men with symptomatic testosterone deficiency identified at Men's Health Boston (MHB), an outpatient men's health clinic.

In a pilot study involving 32 blood samples, investigators have already identified a specific metabolomic signature in men undergoing androgen deprivation therapy for prostate cancer. Based on these preliminary results and other recent studies, investigators hypothesize that they can detect metabolic derangements in men with T deficiency and that these derangements will respond to changes in T levels. Investigators will address this hypothesis though the following specific aims:

Aim 1: To characterize metabolite profiles and evaluate metabolic dysfunction in T deficient men

To accomplish this aim investigators will study T deficient men presenting to MHB. In addition to metabolite profiling, these men will undergo a comprehensive clinical evaluation at MHB including:

* Complete History and Physical exam
* Assessment of symptoms of T deficiency and sexual function using validated and other questionnaires
* Comprehensive hormonal and metabolic laboratory evaluation
* Body composition (including visceral and subcutaneous adiposity) by dual x-ray absorptiometry (DXA) Investigators will build a reference dataset relating metabolite profiles with metabolic risk factors in a clinical population of T deficient men. This will include data on the relationship between metabolite profiles and sexual and other symptoms of T deficiency. Investigators will also compare concentrations of select metabolites between T deficient men and matched eugonadal controls previously studied in the Framingham cohort.

Aim 2: To determine how T therapy influences metabolite profiles and IR

1. To identify metabolites that change in response to raising serum T
2. To determine how changes in metabolite profiles relate to changes in IR
3. To determine how response in terms of sexual function symptoms of low T relate to response in metabolite profiles and IR.

Metabolite profiles will be obtained and clinical evaluation performed (described above under Aim1) at baseline and again after 6 months of therapy. Investigators will study interactions between changes in sexual function and serum T, IR, body composition and metabolite profiles (with particular attention to established metabolite markers of IR).

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic testosterone deficiency
* Intend to undergo testosterone therapy at Men's Health Boston
* Total testosterone <350ng/dL or free testosterone <1.5ng/dL

Exclusion Criteria:

* Type 1 diabetes
* Use of exogenous testosterone or clomiphene citrate
* Known karyotype abnormalities
* Seizure disorders
* Malignancy

Ages: 20 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Testosterone deficient men who intend to undergo testosterone therapy at an outpatient men's health clinic.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-07; Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Metabolomics | After 4-6 mo of therapy
  Blood samples will be sent to the Metabolite Profiling Platform at the Broad Institute of Harvard/Massachusetts Institute of Technology. Metabolomics measures hundreds of unique chemical markers (metabolites) involved in normal and diseased cellular processes from a blood sample. These metabolites include branched chain and aromatic amino acids, ketoacids, and triacylglycerides.
Metabolomics | Baseline
  Blood samples will be sent to the Metabolite Profiling Platform at the Broad Institute of Harvard/Massachusetts Institute of Technology. Metabolomics measures hundreds of unique chemical markers (metabolites) involved in normal and diseased cellular processes from a blood sample. These metabolites include branched chain and aromatic amino acids, ketoacids, and triacylglycerides.

SECONDARY OUTCOMES:
Symptoms of Testosterone Deficiency | After 4-6mo of T therapy
  Symptoms of T deficiency will be assessed using the clinical history and using validated and other questionnaires.
Body Composition | After 4-6mo of T therapy
  Body composition, including visceral and subcutaneous adiposity, will be determined using dual energy x-ray absorptiometry (DXA)
Fasting insulin and glucose | After 4-6mo of T therapy
  Insulin and glucose will be determined from a fasting blood sample.
Lipid Profile | After 4-6mo of T therapy
  A clinical lipid profile including LDL, HDL, and total triglycerides will be obtained from a fasting blood sample.
Symptoms of Testosterone Deficiency | Baseline
  Symptoms of T deficiency will be assessed using the clinical history and using validated and other questionnaires.
Body Composition | Baseline
  Body composition, including visceral and subcutaneous adiposity, will be determined using dual energy x-ray absorptiometry (DXA)
Fasting insulin and glucose | Baseline
  Insulin and glucose will be determined from a fasting blood sample.
Lipid Profile | Baseline
  A clinical lipid profile including LDL, HDL, and total triglycerides will be obtained from a fasting blood sample.

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Morgentaler, MD, Principal Investigator — Men's Health Boston; Ravi Kacker, MD, Study Director — Men's Health Boston
Locations (1):
- Men's Health Boston, Chestnut Hill, Massachusetts, United States

REFERENCES:
- [Background] Cheng S, Rhee EP, Larson MG, Lewis GD, McCabe EL, Shen D, Palma MJ, Roberts LD, Dejam A, Souza AL, Deik AA, Magnusson M, Fox CS, O'Donnell CJ, Vasan RS, Melander O, Clish CB, Gerszten RE, Wang TJ. Metabolite profiling identifies pathways associated with metabolic risk in humans. Circulation. 2012 May 8;125(18):2222-31. doi: 10.1161/CIRCULATIONAHA.111.067827. Epub 2012 Apr 11. PMID 22496159
- [Background] Wang TJ, Larson MG, Vasan RS, Cheng S, Rhee EP, McCabe E, Lewis GD, Fox CS, Jacques PF, Fernandez C, O'Donnell CJ, Carr SA, Mootha VK, Florez JC, Souza A, Melander O, Clish CB, Gerszten RE. Metabolite profiles and the risk of developing diabetes. Nat Med. 2011 Apr;17(4):448-53. doi: 10.1038/nm.2307. Epub 2011 Mar 20. PMID 21423183
- [Background] Rhee EP, Cheng S, Larson MG, Walford GA, Lewis GD, McCabe E, Yang E, Farrell L, Fox CS, O'Donnell CJ, Carr SA, Vasan RS, Florez JC, Clish CB, Wang TJ, Gerszten RE. Lipid profiling identifies a triacylglycerol signature of insulin resistance and improves diabetes prediction in humans. J Clin Invest. 2011 Apr;121(4):1402-11. doi: 10.1172/JCI44442. Epub 2011 Mar 14. PMID 21403394
- [Background] Kapoor D, Goodwin E, Channer KS, Jones TH. Testosterone replacement therapy improves insulin resistance, glycaemic control, visceral adiposity and hypercholesterolaemia in hypogonadal men with type 2 diabetes. Eur J Endocrinol. 2006 Jun;154(6):899-906. doi: 10.1530/eje.1.02166. PMID 16728551
- [Background] Heufelder AE, Saad F, Bunck MC, Gooren L. Fifty-two-week treatment with diet and exercise plus transdermal testosterone reverses the metabolic syndrome and improves glycemic control in men with newly diagnosed type 2 diabetes and subnormal plasma testosterone. J Androl. 2009 Nov-Dec;30(6):726-33. doi: 10.2164/jandrol.108.007005. Epub 2009 Jul 3. PMID 19578132